CLINICAL TRIAL: NCT04302272
Title: The Spiration® Valve System (SVS) Post-Market Registry Study for Severe Emphysema
Brief Title: STRIVE Post-Market Registry Study
Status: Recruiting | Type: Observational
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Other Study IDs: 17
Record Dates: First submitted 2020-02-24; First posted 2020-03-10 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Emphysema
Keywords: Emphysema; Chronic obstructive pulmonary disease (COPD); Spiration valve system
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Spiration Valve System (SVS) — Spiration Valves are one-way endobronchial valves indicated for adult patients with shortness of breath and hyperinflation associated with severe emphysema in regions of the lung that have evidence of low collateral ventilation. The Spiration Valve is loaded in the deployment catheter, then passed through the channel of a flexible bronchoscope and deployed at the intended target location. The SVS device is designed to relieve the symptoms of shortness of breath and hyperinflation associated with severe emphysema without surgery.

SUMMARY:
This is a single-arm, prospective, multi-center, Registry study to evaluate the long-term safety and effectiveness of the Spiration Valve System (SVS) for the treatment of severe emphysema in a post-market setting.

DETAILED DESCRIPTION:
This post-market study is a single-arm, prospective, multi-center Registry. It is designed to assess 36-month safety and effectiveness of this FDA approved product in a post-approval setting, and to support the continued assessment of Spiration Valve System therapy for the treatment of severe emphysema in the United States.

Subjects who are eligible and consent to be in this study, will be monitored for outcome data from baseline through 3 years post-first implant.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with shortness of breath and hyperinflation associated with severe emphysema and evidence of low collateral ventilation.
2. Subjects must understand and voluntarily sign an informed consent form.

Exclusion Criteria:

1. Subjects who are not appropriate for SVS therapy based upon the US FDA-approved IFU requirements.
2. Subjects who were withdrawn from this study for any reason will not be allowed to re-enroll.
3. Subjects who have incomplete screening or baseline data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with shortness of breath and hyperinflation associated with severe emphysema in regions of the lung that have evidence of low collateral ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-09 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of pre-specified thoracic adverse events of special interest (TAEsSI) through 12 months following the first implantation procedure | 12 months
  The primary safety endpoint will be the incidence of device-related and procedure-related pre-specified thoracic adverse events of special interest (TAEsSI) through 12 months following the first implantation procedure.
Rate (per patient-year) of pre-specified thoracic adverse events of special interest (TAEsSI) through 36 months following the first implantation procedure | 36 months
  An additional analysis will present the rate (per patient-year) of TAEsSI.

SECONDARY OUTCOMES:
45-day pneumothorax rate | 45 days
  45-day pneumothorax rate, defined as pneumothorax requiring surgical intervention, or prolonged air leak > 7 days defined as the time from chest tube insertion to the time the air leak is not present.
Survival rate over 24 months | 24 months
  Survival rate over 24 months compared to the EMPROVE study control cohort

OTHER OUTCOMES:
Targeted lobe volume reduction (TLVR) | 6 months
  Target lobe volume reduction (TLVR) determined from quantitative High-Resolution Computed Tomography (HRCT) at 6 months
Hyperinflation | 6 and 12 months
  It will be measured by the ratio of residual volume to total lung capacity (RV/TLC) using plethysmography from baseline
Forced expiratory volume in 1 second (FEV1) | 6, 12, 24 and 36 months
  Relative (percentage) change from baseline at 6, 12, 24 and 36 months
Modified Medical Research Council (mMRC) change | 6, 12, 24 and 36 months
  Modified Medical Research Council (mMRC) change from baseline at 6, 12, 24 and 36 months
St. George's Respiratory Questionnaire (SGRQ) change | 6, 12, 24 and 36 months
  St. George's Respiratory Questionnaire (SGRQ) change from baseline at 6, 12, 24 and 36 months
6 Minute Walk Test (6MWT) change | 6 and 12 months
  6-minute walk test (6MWT) change from baseline at 6 and 12 months
Body Mass, Airflow Obstruction, Dyspnea and Exercise Capacity (BODE) Index change | 6 and 12 months
  Body mass, Airflow Obstruction, Dyspnea and Exercise Capacity (BODE) Index change from baseline at 6 and 12 months
Responder Rates based on Minimum Clinically Important Difference (MCID) | 3 years
  Responder rates based on Minimum Clinically Important Difference (MCID) for Effectiveness Observations

CONTACTS AND LOCATIONS:
Overall Officials: Gerard Criner, MD, Principal Investigator — Temple University
Locations (13):
- United States (13):
  - Dignity Health St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - El Camino, Taft Center for Clinical Research, Mountain View, California
  - Northwestern University, Division of Pulmonary and Critical Care Medicine, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - LSU Health Shreveport, Shreveport, Louisiana
  - Beth Israel Decaconess, Boston, Massachusetts
  - Memorial Hospital at Gulfport, Gulfport, Mississippi
  - Duke University Medical Center, Durham, North Carolina
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - Baylor Scott & White Research Institute, Dallas, Texas
  - University of Texas Southwestern, Dallas, Texas